CLINICAL TRIAL: NCT05853133
Title: Evaluation of Postoperative Quality of Recovery Score in Radical Prostatectomy Cases With Erector Spinae Plane Block and Wound Infiltration
Brief Title: Evaluation of Postoperative Quality of Recovery Score in Radical Prostatectomy With Erector Spinae Plane Block
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Eskisehir Osmangazi University (Other)
Responsible Party: Principal Investigator, Meryem Onay, Assistant Professor-Anesthesiologist, Eskisehir Osmangazi University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ESOGU 5
Record Dates: First submitted 2023-05-02; First posted 2023-05-10 (Actual); Last update posted 2024-02-13 (Actual); Status verified 2024-02

CONDITIONS: Postoperative Pain
Keywords: Erector Spinae Plane Block; Wound Infiltration; Radical Prostatectomy; Postoperative Pain
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Intervention Model Description: Group E: Before the operation, the ESP block will be applied to the patients bilaterally, in the prone position under sedation by same anesthesiologist. Group E (ESP block) will be applied 20 ml of %0.25 bupivacaine between the erector spina muscle and transverse process at the 11th thoracic level.
  Group W: At the end of the operation,wound infiltration will be administered under general anesthesia in supine position by surgeon. Subfascial and subcutaneous wound infiltration is performed (20 ml of 0.25% bupivacaine each)
  In the postoperative period, the patient was evaluated to the groups at the 2st and 6th, 12th and 24th hours. Visual pain scores (VAS) in rest and movement, hemodynamic values, tramadol consumption, nausea-vomiting score, ramsey sedation scale, postoperative complications will be recorded. A 40-item recovery of quality of score will be applied in the preoperative and postoperative period to evaluate the patient's quality of life.
Who Masked: Investigator, Outcomes Assessor
Masking Description: In the postoperative period, the effectiveness and safety of the block will be evaluated by another researcher (blind) who does not know which group the patient is in.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group E (Active Comparator): ESP block will be applied bilaterally, 20 ml of %0.25 bupivacaine between the erector spinae muscle and transverse process at the 11th thoracic level.
  Interventions: Other: Erector Spinae Plane Block
- Group W (Active Comparator): Subfascial and subcutaneous wound infiltration is performed (20 ml of 0.25% bupivacaine each).
  Interventions: Other: Wound Infiltration

INTERVENTIONS:
Other: Erector Spinae Plane Block — Group E (ESP block), before the operation, the ESP block will be applied to the patients in the prone position under sedation by same anesthesiologist. ESP block will be applied bilaterally, 20 ml of %0.25 bupivacaine between the erector spinae muscle and transverse process at the 11th thoracic level. All patients will be equipped with an IV tramadol patient-controlled analgesia (PCA) device. In the postoperative period, the patient was evaluated by another researcher who blind to the groups at the 2st and 6th, 12th and 24th hours. Visual pain scores (VAS) in rest and movement, hemodynamic values, tramadol consumption, nausea-vomiting score, ramsey sedation scale, postoperative complications will be recorded. A 40-item recovery of quality of score will be applied in the preoperative and postoperative period to evaluate the patient's quality of life.
  Other Names: Group E
  Arms: Group E
Other: Wound Infiltration — Group W, at the end of the operation,wound infiltration will be administered under general anesthesia in supine position by same surgeon. Subfascial and subcutaneous wound infiltration is performed (20 ml of 0.25% bupivacaine each). All patients will be equipped with an IV tramadol patient-controlled analgesia (PCA) device. In the postoperative period, the patient was evaluated by another researcher who blind to the groups at the 2st and 6th, 12th and 24th hours. Visual pain scores (VAS) in rest and movement, hemodynamic values, tramadol consumption, nausea-vomiting score, ramsey sedation scale, postoperative complications will be recorded. A 40-item recovery of quality of score will be applied in the preoperative and postoperative period to evaluate the patient's quality of life.
  Other Names: Group W
  Arms: Group W

SUMMARY:
Radical prostatectomy is performed with a median incision below the umbilicus. Although the position is supine, the waist extension movement is created in order to facilitate access to the surgical site. The investigator think that this may be a factor affecting the postoperative comfort, not only in the pain in the surgical field, but especially in patients with low back pain (facet joint pain, etc.). Techniques that provide quality postoperative recovery with reduced morbidity and rapid return to daily activities are important for anesthesiologists.

In this study, the investigator aimed to evaluate the postoperative recovery quality (Quality of Recovery score (QoR-40)) of patients who underwent open radical prostatectomy and underwent erector spina plan block and wound infiltration for postoperative analgesia.

DETAILED DESCRIPTION:
Patients will be randomly divided into 2 groups as Group E (ESP block) and Group W (Wound Infiltration). Before the operation, the ESP block will be applied to the patients in the prone position under sedation by same anesthesiologist. Group E (ESP block) will be applied bilaterally, 20 ml of %0.25 bupivacaine between the erector spinae muscle and transverse process at the 11th thoracic level. Fifteen minutes after the block, the patient's dermotamal examination will be evaluated and patients with successful block will be included in the study.At the end of the operation,wound infiltration will be administered under general anesthesia in supine position by surgeon. Subfascial and subcutaneous wound infiltration is performed (20 ml of 0.25% bupivacaine each). At the end of the operation, the patients with a Modified aldreate score ≥9 will be sent from the postoperative anesthesia unit. All patients will be equipped with IV tramadol patient-controlled analgesia (PCA) device. The solution will be prepared such that tramadol is 4 mg / ml. PCA 10 mg bolus dose will be delivered with 15 min lock-out time. In the postoperative period, the patient was evaluated by another researcher who blind to the groups at the 2st and 6th, 12th and 24th hours. Visual pain scores (VAS) in rest and movement, hemodynamic values, tramadol consumption, nausea-vomiting score, ramsey sedation scale, postoperative complications will be recorded. A 40-item recovery of quality of score will be applied in the preoperative and postoperative period to evaluate the patient's quality of life.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologist physical status I-III
* Radical prostatectomy

Exclusion Criteria:

* Infection in the incision area
* Coagulation disorder
* Known allergy history against to the study drugs
* Lack of adequate cognitive activity in the use of patient-controlled analgesia and VAS

Ages: 18 Years to 70 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — radical prostatectomy surgery
Enrollment: 52 (Actual)
Dates: Start 2023-05-16 (Actual); Primary Completion 2024-02-01 (Actual); Study Completion 2024-02-04 (Actual)

PRIMARY OUTCOMES:
Postoperative Quality Of Recovery Score in Radical Prostatectomy | Postoperative 24 hours
  QoR-40, a 40-item questionnaire that provides a global score and subscores across five dimensions: patient support, comfort, emotions, physical independence, and pain. Each item is rated on a scale of 1-5, providing a minimum score of 40 and maximum of 200. The QoR-40 scores range from 40 to 200 with a 200 representing a better recovery outcome

SECONDARY OUTCOMES:
Total opiate consumption | 24 hours
  Total tramadol patient control analgesia prepared 4 mg / ml. PCA 10 mg bolus dose will be delivered with 15 min lock-out time. Follow up tramadol consumption at postoperative 24 hours
postoperative pain scores | 24 hours
  Visual analog scale at rest and movement (0 (no pain)-10 (unbearable pain))

CONTACTS AND LOCATIONS:
Overall Officials: Meryem Onay, Principal Investigator — Eskisehir Osmangazi University Faculty Of Medıcıne
Locations (1):
- Eskisehir Osmangazi University Faculty of Medicine, Eskişehir, Odunpazarı, Turkey (Türkiye)

REFERENCES:
- [Background] Elkassabany N, Ahmed M, Malkowicz SB, Heitjan DF, Isserman JA, Ochroch EA. Comparison between the analgesic efficacy of transversus abdominis plane (TAP) block and placebo in open retropubic radical prostatectomy: a prospective, randomized, double-blinded study. J Clin Anesth. 2013 Sep;25(6):459-65. doi: 10.1016/j.jclinane.2013.04.009. Epub 2013 Aug 17. PMID 23965191
- [Background] Dost B, Kaya C, Ozdemir E, Ustun YB, Koksal E, Bilgin S, Bostanci Y. Ultrasound-guided erector spinae plane block for postoperative analgesia in patients undergoing open radical prostatectomy: A randomized, placebo-controlled trial. J Clin Anesth. 2021 Sep;72:110277. doi: 10.1016/j.jclinane.2021.110277. Epub 2021 Apr 7. PMID 33838536
- [Background] Tulgar S, Senturk O. Ultrasound guided low thoracic erector spinae plane block for postoperative analgesia in radical retropubic prostatectomy, a new indication. J Clin Anesth. 2018 Jun;47:4. doi: 10.1016/j.jclinane.2018.02.013. Epub 2018 Mar 5. No abstract available. PMID 29518667
- [Background] Osaheni O, Idehen HO, Imarengiaye CO. Analgesia for postoperative myomectomy pain: A comparison of ultrasound-guided transversus abdominis plane block and wound infiltration. Niger J Clin Pract. 2020 Nov;23(11):1523-1529. doi: 10.4103/njcp.njcp_162_19. PMID 33221776
- [Background] Lemoine A, Witdouck A, Beloeil H, Bonnet F; PROSPECT Working Group Of The European Society Of Regional Anaesthesia And Pain Therapy (ESRA). PROSPECT guidelines update for evidence-based pain management after prostatectomy for cancer. Anaesth Crit Care Pain Med. 2021 Aug;40(4):100922. doi: 10.1016/j.accpm.2021.100922. Epub 2021 Jun 29. PMID 34197976
- [Background] Canitez A, Kozanhan B, Aksoy N, Yildiz M, Tutar MS. Effect of erector spinae plane block on the postoperative quality of recovery after laparoscopic cholecystectomy: a prospective double-blind study. Br J Anaesth. 2021 Oct;127(4):629-635. doi: 10.1016/j.bja.2021.06.030. Epub 2021 Jul 31. PMID 34340839
- [Background] Myles PS, Weitkamp B, Jones K, Melick J, Hensen S. Validity and reliability of a postoperative quality of recovery score: the QoR-40. Br J Anaesth. 2000 Jan;84(1):11-5. doi: 10.1093/oxfordjournals.bja.a013366. PMID 10740540